CLINICAL TRIAL: NCT04956614
Title: Comparison of Therapeutic Effect of Different Brace Fixed Time After Novel Achilles Tendon Rupture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM2020252
Record Dates: First submitted 2021-07-02; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Achilles Tendon Rupture
Keywords: Duration of immobilisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suture of Achilles tendon without immobilisation (Experimental)
  Interventions: Device: immobilisation duration
- suture of Achilles tendon with immobilisation (Experimental)
  Interventions: Device: immobilisation duration

INTERVENTIONS:
Device: immobilisation duration — immobilisation duration of 2,4,6 week after suture of Achilles tendon

SUMMARY:
This study is a prospective randomized controlled clinical study. After the novel Achilles tendon rupture repaired , patients were randomly divided into 4 groups according to immobilisation duration of 0, 2, 4, and 6 weeks, respectively. All patients underwent the same suture technique with a similar rehabilitation protocol and were examined clinically at 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks to study the difference in efficacy among the groups.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical study is designed to compare the treatment outcomes of different immobilisation duration by dividing the patients into four groups according to immobilisation duration of 0, 2, 4, and 6 weeks after a similar suture technique. The primary outcome was the time of return to light sports activity (LSA). Secondary outcomes included range of motion (ROM) and single-legged heel rise height (SHRH). Data on operation time, complications, visual analogue pain scale (VAS), American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score, and Achilles tendon Total Rupture score (ATRS) were also collected. Demographic baseline data were analysed using one-way analysis of variance; outcome parameters were analysed using Kruskal-Wallis H test, and complications were analysed using Fisher's exact test. Statistical significance was considered at P ≤ 0.05.

The inclusion criteria were patients aged 18 to 60 years with an acute closed single-legged complete ATR who underwent open surgery with our suture technique.

The excluded criteria were patients with prior ATR and those without rehabilitation or follow-up outcomes. Other situations that affected patients' lower limb functions or tendon healing (e.g. autoimmune disease, diabetes mellitus, systemic corticosteroid treatment) were also excluded.

ELIGIBILITY:
Inclusion Criteria:

patients aged 18 to 60 years with an acute closed single-legged complete ATR who underwent open surgery with our suture technique.

Exclusion Criteria:

* patients with prior Achilles tendon rupture or other situations that affected their lower limb functions or tendon healing (e.g., autoimmune disease, diabetes mellitus, systemic corticosteroid treatment).

  * an inability to complete our suture technique (e.g., the distance from the rupture site to the Achilles tendon insertion was less than 3.5 cm) .
  * those without rehabilitation or follow-up outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
The time of return to light sports activity | From operation to 1-year follow-up after the surgery
  When the patients are able to do jogging or rapid walk after the surgery, the time will be recorded

SECONDARY OUTCOMES:
Range of motion (ROM) recovery time | From operation to 1-year follow-up after the surgery
  The recovery time will be recorded when the ROM is similar to that of the uninjured side.
Recovery time of the single-legged heel rise height (SHRH) | From operation to 1-year follow-up after the surgery
  The heel rise height is measured as the distance from the ground to the heel when the patient lift the heel while keeping the knee straight. The recovery time is noted when the SHRH is similar to that of the opposite leg.

OTHER OUTCOMES:
visual analogue scale (VAS) | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  VAS pain score is from 0 to 10, the higher score demonstrate the more severe pain.
  VAS pain score is from 0 to 10, the higher score demonstrate the more severe pain.
American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  The AOFAS score ranges from 0 to 100, with a healthy hindfoot receiving 100 points.
the Achilles tendon Total Rupture Score (ATRS) | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  The ATRS includes 10 items; each item has a score ranging between 0 and 10 on a Likert scale, with 100 indicating no major limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No